CLINICAL TRIAL: NCT03400163
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multiple Dose Sub-study to Evaluate the Safety, Pharmacokinetics and Pharmacodynamic Effects of BMS-986036 in Adults With Non-alcoholic Steatohepatitis
Brief Title: A Sub-study of BMS-986036 in Subjects With Non-Alcoholic Steatohepatitis (NASH)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MB130-045 A
Record Dates: First submitted 2018-01-02; First posted 2018-01-17 (Actual); Results first posted 2020-02-19 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Non-Alcoholic Steatohepatitis
Keywords: First Line Therapy; NASH
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Pegbelfermin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group D: (Experimental): Administered as specified on specified days
  Interventions: Drug: BMS-986036
- Treatment Group E: (Placebo Comparator): Administered as specified on specified days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BMS-986036 — BMS-986036 20 mg QD
  Arms: Treatment Group D:
Drug: Placebo — Placebo QD
  Arms: Treatment Group E:

SUMMARY:
The purpose of this sub-study of MB130-045 is to determine the pharmacokinetic effects, pharmacodynamic effects, efficacy and safety of BMS-986036 20 mg QD in subjects with Non-alcoholic Steatohepatitis (NASH)

ELIGIBILITY:
For more information regarding BMS clinical trial participation, please visit www.BMSStudyConnect.com

Inclusion Criteria:

* Male or female between 21 and 75 years old
* Body Mass Index (BMI) of 25 or more

Exclusion Criteria:

* Chronic Liver disease other than NASH
* Uncontrolled diabetes
* Any major surgery within 6 weeks of screening
* Unable to self-administer under the skin injections
* Any bone trauma, fracture or bone surgery within 8 weeks of screening

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2015-05-08 (Actual); Primary Completion 2017-01-18 (Actual); Study Completion 2017-06-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (2):
- United States (2):
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Texas Liver Institute, San Antonio, Texas

REFERENCES:
- See also: BMS Clinical Trial Patient Recruiting — http://bms.com/studyconnect/Pages/home.aspx
- See also: Investigator Inquiry Form — http://www.bms.com/clinical_trials/Pages/Investigator_inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 participants were enrolled, randomized and treated within this sub-study (PK cohort).
  Note: parent study is NCT02413372 (MB130-045).
Groups:
- BMS-986036 20 mg QD: Participants self-administered 20 mg subcutaneous (SC) injections of BMS-986036, once daily (QD), for 16 weeks in a double-blind, outpatient setting
- Placebo 20 mg QD: Participants self-administered SC injections of placebo, once daily, for 16 weeks in a double-blind, outpatient setting.
Period: Treatment Period
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0
Period: Follow-up Period
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Started | 1 | 2
Completed | 1 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD | Total
Number analyzed (Participants) | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35 (NA) — only 1 participant within category | 49.5 (2.12) | 44.67 (8.50)
Age, Customized [Count of Participants; unit: Participants] — Age categorization
  Participants
    < 65 years of age | 1 | 2 | 3
    >= 65 years of age | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 2
  Not Hispanic or Latino | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 2 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in Percent Hepatic Fat Fraction (%) by Magnetic Resonance Imaging (MRI) From Baseline to Week 16
Description: The mean change in percent hepatic fat fraction (%) by MRI from baseline to Week 16 was assessed for each arm. A longitudinal repeated measures analysis was used to analyze the change in hepatic fat fraction (%) at Week 16 from baseline in the treated population who have both a baseline and at least one post-baseline measurement.
Time Frame: From Day 1 to Day 112
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Mean (90% Confidence Interval); unit: percentage
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
percentage | NA [NA to NA] — data not reported due to privacy reasons | NA [NA to NA] — data not reported due to privacy reasons

2. Primary Outcome: Number of Participants With Adverse Events (AEs)
Description: The number of participants with on-study AEs was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Number; unit: Participants
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Participants | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons

3. Primary Outcome: Number of Participants With Serious Adverse Events (SAEs)
Description: The number of participants with on-study SAEs was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Number; unit: Participants
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Participants | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons

4. Primary Outcome: Number of Participants With Injection Site Reactions
Description: The number of participants with on-study injection site reactions was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Number; unit: Participants
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Participants
  Injection Site Bruising | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons
  Injection Site Erythema | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons
  Injection Site Reaction | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons
  Injection Site Pain | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons
  Injection Site Rash | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons
  Injection Site Swelling | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons

5. Primary Outcome: Number of Participants With Adverse Events Leading to Discontinuation
Description: The number of participants with on-study AEs leading to discontinuation was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Number; unit: Participants
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Participants | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons

6. Primary Outcome: Number of Deaths
Description: The number of deaths was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Number; unit: Participants
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Participants | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons

7. Primary Outcome: Number of Participants With Marked Laboratory Abnormalities
Description: The number of participants whose worst toxicity grade increased from baseline to grade 3 or 4 (Toxicity Scale: DAIDS Version 1.0) is reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Number; unit: Participants
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Participants
  Alanine Aminotransferase (ALT) | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons
  Glucose, Fasting - high | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons

8. Primary Outcome: Number of Participants With Vital Sign Abnormalities
Description: The number of participants with out-of-range vital signs noted during interim or final vital sign assessments was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Number; unit: Participants
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Participants | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons

9. Primary Outcome: Number of Participants With Electrocardiogram (ECG) Abnormalities
Description: The number of participants with out-of-range ECG intervals observed during interim or final electrocardiogram assessments was reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Number; unit: Participants
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Participants
  PR > 200 msec | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons
  QRS > 120 msec | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons
  QT > 500 msec | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons
  QTcF > 450 msec | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons
  QT change from baseline > 30 msec | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons
  QTcF change from baseline > 30 msec | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons

10. Primary Outcome: Number of Participants With Physical Examination Abnormalities
Description: The number of participants with abnormalities observed during interim or final physical examination assessments is reported for each arm.
Time Frame: From first dose to date of last dose plus 30 days
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Number; unit: Participants
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Participants | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons

11. Primary Outcome: Mean Percent Change From Baseline in Bone Mineral Density by Dual Energy X-Ray Absorptiometry (DXA)
Description: The mean percent change in bone mineral density from baseline to day 112 reported for each arm.
Time Frame: From Day 1 to Day 112
Population: All treated participants with DXA data at baseline and 6 months
  Note: data not reported due to privacy reasons
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Percentage | NA (NA) — data not reported due to privacy reasons | NA (NA) — data not reported due to privacy reasons

12. Secondary Outcome: Geometric Mean of Trough Observed Plasma Concentration (Ctrough) of BMS-986036 at Day 112
Description: The observed serum concentration of BMS-986036 before the next dose is administered (pre-dose concentration) was assessed for both C-terminal intact and total molecule. Geometric means are presented for each arm.
Time Frame: From Day 1 to Day 112
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
ng/mL
  C-Terminal Intact | NA (NA) — data not reported due to privacy reasons | NA (NA) — data not reported due to privacy reasons
  Total | NA (NA) — data not reported due to privacy reasons | NA (NA) — data not reported due to privacy reasons

13. Secondary Outcome: Number of Participants With Positive Anti-BMS-986036 Antibody (ADA) Response at Day 142
Description: Participants were monitored for antibodies to study medication using a validated ADA homogenous bridge assay with BMS-986036 and electrochemical luminescence detection. The number of treated participants with positive Anti-BMS-986036 antibody titers up to Day 142 with regards to baseline was reported for each arm.
Time Frame: From Day 1 to Day 142
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Number; unit: Participants
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Participants | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons

14. Secondary Outcome: Number of Participants With Positive Anti-FGF21 Antibody Response at Day 142
Description: Participants were monitored for antibodies to FGF21 using a validated homogenous bridge assay with Met-FGF21 (recombinant produced) and electrochemical luminescence detection. The number of treated participants with positive Anti-FGF21 antibody titers up to Day 142 with regards to baseline was reported for each arm.
Time Frame: From Day 1 to Day 142
Population: All treated participants
  Note: data not reported due to privacy reasons
Measure: Number; unit: Participants
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
Number analyzed (Participants) | 1 | 2
Participants | NA — data not reported due to privacy reasons | NA — data not reported due to privacy reasons

ADVERSE EVENTS:
Time Frame: Non-serious adverse events after first dose of study medication and within 7 days of last dose and serious adverse events after first dose of study medication and within 30 days of last dose (approximately 4 months).
Description: data not reported due to privacy reasons
Arm/Group | BMS-986036 20 mg QD | Placebo 20 mg QD
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2016-06-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT03400163/Prot_000.pdf
  • Statistical Analysis Plan (2017-09-18): https://cdn.clinicaltrials.gov/large-docs/63/NCT03400163/SAP_001.pdf